CLINICAL TRIAL: NCT00835289
Title: The Chronic Obstructive Pulmonary Disease Fish Oil Pilot Trial
Acronym: COD-Fish
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: National Institute of Environmental Health Sciences (NIEHS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AAAC9586; P30ES009089 (NIH)
Record Dates: First submitted 2008-10-22; First posted 2009-02-03 (Estimated); Last update posted 2020-11-17 (Actual); Status verified 2020-11

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Clinical Trials, Randomized
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Fatty Acids, Omega-3; Docosahexaenoic Acids

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (corn oil) (Placebo Comparator): Each participant will be taking 3 capsules of a matching placebo (corn oil).
  Interventions: Other: Placebo
- PUFA (Omax3) (Experimental): Omax3[TM] (Cenestra Health), or dietary supplement: n-3 polyunsaturated fatty acids, is a 1 gram softgel capsule containing 94.5% omega-3 fatty acids. Each participant will be taking 3 capsules of Omax3[TM].
  Interventions: Dietary Supplement: n-3 polyunsaturated fatty acids

INTERVENTIONS:
Dietary Supplement: n-3 polyunsaturated fatty acids — Omax3[TM] (Cenestra Health [TM]) is a 1 g softgel capsule containing 94.5% omega-3 fatty acids. Each serving size is a 1 gram capsule, which contains 690 mg of eicosapentanoic acid (EPA) and 182 mg of docosahexanoic acid (DHA). Inactive ingredients include: Vitamin E/Tocopherol 2294 ppm (in a carrier of partially hydrogenated vegetable oils including soybean oil), gelatin, glycerol, and purified water (components of the capsule shell). The study participants will be randomized to 3 softgel capsules a day for 6 months.
  Other Names: Omax-3; PUFA; Omega-3
  Arms: PUFA (Omax3)
Other: Placebo — 3 capsules of matching corn oil placebo
  Arms: Placebo (corn oil)

SUMMARY:
Chronic obstructive pulmonary disease (COPD) is currently the fourth leading cause of death in the United States. Unlike the other leading causes of death, no medical therapies currently available improve the course of disease or affect survival in COPD. Recent investigations suggest that endothelial dysfunction and chronic inflammation is fundamental to COPD. Fish oil intake improves endothelial dysfunction and lowers levels of inflammatory intermediaries which may be important in the development of COPD.

The Chronic Obstructive Pulmonary Disease Fish Oil (COD-Fish) Pilot Trial will enroll 40-45 participants with COPD. These participants will be randomized to receive omega-3 polyunsaturated fatty acid supplementation (PUFA) or placebo (containing corn oil). All participants will perform a number of noninvasive tests (including flow-mediated dilation (FMD) and pulmonary function testing) at study entry as well as every two months for a total of six months. Thirty participants who agree to it will undergo a separate procedure to collect cells from inside a forearm vein for analysis to be compared to 30 controls. The main purpose of this trial is to examine the effect of PUFA on endothelial function as measured by change in FMD in patients with COPD. We hypothesize that in subjects with COPD, treatment with PUFA will increase FMD.

DETAILED DESCRIPTION:
Chronic obstructive pulmonary disease is abbreviated as COPD and includes both emphysema and chronic bronchitis. COPD is currently the fourth leading cause of death in the United States. Unlike most major medical diseases, the morbidity and mortality from COPD continue to rise in the US. In 2000, over 10 million Americans carried a physician diagnosis of COPD and 120,000 Americans died from this disease. Additionally, from the year 1980 to the year 2000, the number of cases of COPD among women nearly doubled and the prevalence among African Americans increased by 61%. Unlike the other leading causes of death, no medical therapies currently available improve the course of disease or affect survival in COPD. Current therapies for COPD that improve survival in COPD are limited to smoking cessation, oxygen therapy, and possibly surgery. Medical therapies such as inhalers and pills improve symptoms and reduce COPD exacerbations ("attacks"), but have not been shown to slow down the progression of the disease.

Recent investigations suggest that endothelial dysfunction and chronic inflammation is fundamental to COPD. Fish oil intake improves endothelial dysfunction and lowers levels of inflammatory intermediaries. These inflammatory intermediaries can be measured in the blood and are potentially important in the development of COPD. Large observational studies demonstrate that participants who eat high amounts of fish oil develop less COPD and have lower levels of these inflammatory intermediaries.

The Chronic Obstructive Pulmonary Disease Fish Oil (COD-Fish) Pilot Trial will enroll 40-45 participants with COPD. These participants will be randomized to receive Omax3[TM] or placebo (containing corn oil). Omax3[TM] (Cenestra Health) is a 1 gram softgel capsule containing 94.5% omega-3 fatty acids. Each participant will be taking 3 capsules of either Omax3[TM] or matching placebo. The investigators and the subjects will be blinded, meaning that neither the investigators nor the subjects will know if they are taking Omax3[TM] or placebo. All participants will perform a number of noninvasive tests at study entry as well as every two months for a total of six months. They will also undergo pulmonary function testing, flow-mediated dilation (FMD), peripheral arterial tonometry (PAT), six minute-walk tests (6MWT), blood drawing and answer questionnaire data. Thirty participants who agree to it will undergo a separate procedure to collect cells from inside a forearm vein for analysis to be compared to 30 controls. The main purpose of this trial is to examine the effect of Omax3[TM] on endothelial function as measured by change in FMD in patients with COPD. We hypothesize that in subjects with COPD, treatment with Omax3[TM] will increase FMD.

ELIGIBILITY:
Inclusion Criteria:

* Post-bronchodilator FEV1/FVC ratio <70%
* Post-bronchodilator FEV1 <65% predicted.
* Clinical diagnosis of COPD
* Stable medical regimen for 30 days prior to enrollment
* Age > 40 years old
* History of former cigarette smoking, > or = 10 pack years

Exclusion Criteria:

* COPD exacerbation or hospitalization for COPD in the past 30 days
* Confirmed history of physician-diagnosed asthma
* History of unrelated pulmonary disease (e.g. interstitial lung disease, thromboembolic disease)
* Status-post lung transplantation or Lung volume reduction surgery (LVRS)
* Systolic blood pressure >170mmHg or<100mmHg at rest, diastolic blood pressure >100 at rest, or resting HR >120.
* Active cigarette smoking
* Clinical diagnosis of left-sided congestive heart failure
* Clinical diagnosis of coronary artery disease
* Clinical diagnosis of cerebrovascular disease
* Clinical diagnosis of peripheral vascular disease
* Prior history of stroke or myocardial infarction
* Clinical diagnosis of obstructive sleep apnea
* Pregnancy (known, and screen with urine BHCG) or current breastfeeding
* Contraindication to Omax3[TM] use, including a history of hypersensitivity to Omax3[TM]
* Current use of high-dose fish oil capsules (defined as >1 or 2 grams/day of omega-3 fatty acids)
* Current use of Coumadin
* Elevated ALT greater than 2 times the upper limit of normal at baseline
* Congenital abnormality of the arm or hand
* Raynaud's Phenomenon
* History of radical mastectomy or removal or axillary lymph nodes
* Allergy to fish or corn oil
* Unstable angina during previous month
* End Stage Liver Disease, Cirrhosis

For Non-COPD controls (Same Inclusion and exclusion criteria, except for inclusion, must NOT have the following:)

* Post-bronchodilator FEV1/FVC ratio >70%
* Post-bronchodilator FEV1 <65% predicted.
* Clinical diagnosis of COPD

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2009-03; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Percent Flow Mediated Dilation (FMD) | 6 months

SECONDARY OUTCOMES:
Serum level of LTB4 | 6 months
Serum level of TNF-alpha | 6 months
Serum level of IFN-gamma | 6 months
Difference in Pre- and Post-bronchodilator Spirometry | 6 months
Average six-minute-walk test distance | 6 months
Average St. George's Respiratory Questionnaire score | 6 months
Change in percent of Peripheral Arterial Tonometry (EndoPAT) | 4 months
Number of endothelial cell protein expression | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: R Graham Barr, MD/DrPH, Principal Investigator — Columbia University
Locations (1):
- Columbia University Medical Center, New York, New York, United States

REFERENCES:
- [Result] Kim JS, Thomashow MA, Yip NH, Burkart KM, Lo Cascio CM, Shimbo D, Barr RG. Randomization to Omega-3 Fatty Acid Supplementation and Endothelial Function in COPD: The COD-Fish Randomized Controlled Trial. Chronic Obstr Pulm Dis. 2021 Jan;8(1):41-53. doi: 10.15326/jcopdf.8.1.2020.0132. PMID 33150779